CLINICAL TRIAL: NCT02976259
Title: Kinetics of HIV-RNA Decay in Seminal Plasma of Men Receiving a Dolutegravir-based Regimen at the Time of Primary HIV Infection (IMEA 051-DOLUPRIM Study)
Brief Title: Kinetics of HIV-RNA Decay in Seminal Plasma of Men Treated by Dolutegravir at the Time of Primary HIV Infection
Acronym: DOLUPRIM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMEA 051
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-08

CONDITIONS: HIV Infection Primary
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient HIV primary infection (Experimental): HIV primary infection Patient male receiving Dolutegravir
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir — All patients included must have treated by dolutegravir. They will have some exams (plasma samples, sperm samples)

SUMMARY:
Sponsor: IMEA - Fondation Internationale Léon Mba C.H.U. Bichat - Claude Bernard 46, Rue Henri Huchard - 75018 PARIS Tél. : 01.40. 25. 63. 65 - Fax : 01.40.25.63.56

Coordinating investigator:

Dr Caroline Lascoux Combe Hôpital Saint Louis Service Maladies Infectieuses

1 avenue Claude Vellefaux - 75010 PARIS Tél. : 01 42 49 49 73 - Fax : 01 42 49 47 43 E-mail : caroline.lascoux-combe@aphp.fr

Participating country : FRANCE

Primary objective : Comparing the kinetic of HIV-RNA decay in blood plasma and in seminal plasma in patients starting a triple combination regimen with dolutegravir + tenofovir DF (TDF) + emtricitabine (FTC) at the time of PHI.

Secondary objectives :

* Comparison of HIV-1 RNA level in plasma (threshold 20 and 1 copies/ml) and in seminal plasma (threshold 60 copies/ml) at each visit D0, W2, W4, W8, W12, W24, W36, W48
* To assess the frequency of intermittent shedding in seminal plasma once virological suppression has been achieved and until W48
* Evolution of cellular HIV-1 DNA level in PBMC and in non-sperm cells between D0 and W48
* Comparison of dolutegravir concentration in blood plasma and seminal plasma
* Study of risk factors associated with viral persistence of HIV-RNA in the seminal plasma
* Analysis by deep sequencing of the viral population (quasi-species) in both compartments (blood plasma and seminal plasma) before virological suppression has been achieved (i.e. at D0 and W12)

Inclusion criteria :

* Patients diagnosed at the time of primary HIV infection (PHI) (i) a negative or indeterminate HIV ELISA associated with a positive antigenemia or plasma HIV RNA, (ii) a western blot profile compatible with ongoing seroconversion (incomplete western blot with absence of antibodies to pol proteins (p34, p68)) or (iii) an initially negative test for HIV antibodies followed within 3 months by a positive HIV serology
* Treatment including dolutegravir (DTG 50mg) + tenofovir/emtricitabine (TDF/FTC 245 mg/200 mg) initiated by the referee physician within a maximum of 15 days after diagnosis of PHI
* Genotypic sensitivity to TDF, FTC and DTG
* Patient with medical care insurance

Exclusion criteria :

* Chronic infection
* Infection or co-infection with HIV-2

Study treatment : Dolutegravir and tenofovir/emtricitabine Number of subjets : 20 patients (exploratory study)

DETAILED DESCRIPTION:
Secondary objectives :

* Comparison of HIV-1 RNA level in plasma (threshold 20 and 1 copies/ml) and in seminal plasma (threshold 60 copies/ml) at each visit D0, W2, W4, W8, W12, W24, W36, W48
* To assess the frequency of intermittent shedding in seminal plasma once virological suppression has been achieved and until W48
* Evolution of cellular HIV-1 DNA level in PBMC and in non-sperm cells between D0 and W48
* Comparison of dolutegravir concentration in blood plasma and seminal plasma
* Study of risk factors associated with viral persistence of HIV-RNA in the seminal plasma
* Analysis by deep sequencing of the viral population (quasi-species) in both compartments (blood plasma and seminal plasma) before virological suppression has been achieved (i.e. at D0 and W12)

Inclusion criteria :

* Patients diagnosed at the time of primary HIV infection (PHI) (i) a negative or indeterminate HIV ELISA associated with a positive antigenemia or plasma HIV RNA, (ii) a western blot profile compatible with ongoing seroconversion (incomplete western blot with absence of antibodies to pol proteins (p34, p68)) or (iii) an initially negative test for HIV antibodies followed within 3 months by a positive HIV serology
* Treatment including dolutegravir (DTG 50mg) + tenofovir/emtricitabine (TDF/FTC 245 mg/200 mg) initiated by the referee physician within a maximum of 15 days after diagnosis of PHI
* Genotypic sensitivity to TDF, FTC and DTG
* Patient with medical care insurance

Exclusion criteria :

* Chronic infection
* Infection or co-infection with HIV-2

Study treatment : Dolutegravir and tenofovir/emtricitabine Number of subjets : 20 patients (exploratory study)

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed at the time of primary HIV infection (PHI) (i) a negative or indeterminate HIV ELISA associated with a positive antigenemia or plasma HIV RNA, (ii) a western blot profile compatible with ongoing seroconversion (incomplete western blot with absence of antibodies to pol proteins (p34, p68)) or (iii) an initially negative test for HIV antibodies followed within 3 months by a positive HIV serology
* Treatment including dolutegravir (DTG 50mg) + tenofovir/emtricitabine (TDF/FTC 245 mg/200 mg) initiated by the referee physician within a maximum of 15 days after diagnosis of PHI
* Genotypic sensitivity to TDF, FTC and DTG
* Patient with medical care insurance

Exclusion Criteria:

* Chronic infection
* Infection or co-infection with HIV-2

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Comparing the kinetic of HIV-RNA decay in blood plasma and in seminal fluid | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 24 weeks, 36 weeks and 48 weeks
  Measure of HIV-RNA level in blood plasma and seminal fluid at each point and comparaison about the decay between both

SECONDARY OUTCOMES:
The evolution of HIV proviral DNA in the peripheral blood mononuclear cells (PBMC) and in seminal fluid | Day 0 and 48 weeks
Comparison of dolutegravir concentration in blood plasma and seminal fluid | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 24 weeks, 36 weeks and 48 weeks
  Measure of doltegravir concentration in blood and seminal fluid at each points and comparaison of the value between the 2 compartments
Analysis by deep sequencing of the viral population (quasi-species) in both compartments (blood plasma and seminal plasma) before virological suppression has been achieved | Day 0 and 12 weeks

IPD SHARING:
Plan to Share IPD: No